CLINICAL TRIAL: NCT02508025
Title: Towards Better Understanding of FCE Performance in Different Societal Contexts
Acronym: FCEinternat
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Klinik Valens (Other)
Responsible Party: Principal Investigator, Jan Kool, PhD, Klinik Valens
Other Study IDs: EKSG15/079
Record Dates: First submitted 2015-07-21; First posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Musculoskeletal Diseases
Keywords: disability evaluation; psychosocial factors
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Functional Capacity Evaluation — Assessment of work related physical capacity

SUMMARY:
Purposes of this research:

* To study similarities and differences in FCE performances between participants from different countries, jurisdictions, and evaluators.
* To study determinants of FCE performance.

DETAILED DESCRIPTION:
A considerable amount of research has been made on the safety, reliability and validity of the Functional Capacity Evaluation (FCE). Evidence is accumulating on different aspects of validity of FCE in healthy workers and in different patient groups, which has indicated that we are measuring a complex construct consisting of biological, psychological and social variables. However, this knowledge is still unstable as the majority of studies stem from a limited amount of countries. The present project focuses on the biopsychosocial factors that influence FCE performance. Participants undergoing an FCE perform differently depending on biological, psychological and social variables, although the latter has been under-researched. Clinicians are currently unable to predict which factors determine the differences in patient's FCE results. In this project, in addition to biological and psychological variables, investigators include a variety of social variables from different countries, jurisdictions, and evaluators, which may help investigators to identify important determinants of FCE performance. Knowing which characteristics and behaviors are associated with better or poorer participant performances may help clinicians to deliver improved FCE services.

ELIGIBILITY:
Inclusion Criteria:

* Musculoskeletal pain including: back pain, neck pain (including Whiplash-Associated Syndrome grade I or II), upper extremity pain, lower extremity pain.
* Non-specific pain: without specific medical diagnosis, see also exclusion criteria) .
* Complaints' duration > 6 weeks
* Employed or self-employed
* Language skills sufficient to communicate with the FCE-clinician and fill out the required questionnaires

Exclusion Criteria:

* Pregnancy
* Tumours
* Fractures
* Radicular syndromes
* Spondylolisthesis grade 3 or 4)
* Whiplash-Associated Syndrome grade III or IV
* Other specific diagnoses related to the musculoskeletal System
* Unstable cardiovascular conditions and other co-morbidity affecting performance or safety during the FCE (i.e. severe depression needing psychiatric referral).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with non-specific sub-acute or chronic musculoskeletal pain
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Psychological factor: work related fear of movement (minimum 0 - maximum 10) | one day (one measurement only, cross sectional study)
  The fear avoidance beliefs questionnaire has been validated for this purpose
Financial compensation in case of work related disability (% of previous income) | one day (one measurement only, cross sectional study)

SECONDARY OUTCOMES:
Work related physical capacity: max weight safely lifted from floor to waist (kg) | one day (one measurement only, cross sectional study)
  This measure is reliable, safe and valid as it is related to physical work capacity.
Work related physical capacity: distance walked in 6 minutes (meters) | one day (one measurement only, cross sectional study)
  This measure is reliable, safe and valid as it is related to physical work capacity.
Work related physical capacity: grip strength (kg) | one day (one measurement only, cross sectional study)
  This measure is reliable, safe and valid as it is related to physical work capacity.